CLINICAL TRIAL: NCT03019744
Title: Studio Clinico di Efficacia Della Stimolazione Elettrica Funzionale Controllata da Segnale Elettromiografico Nel Trattamento Dell'Arto Superiore in Pazienti Con Esiti di Ictus Cerebrovascolare (Progetto Rises)
Brief Title: Efficacy Study of FES Controlled by Electromyographic Signal for the Treatment of Upper Limb in Post-stroke Patients
Acronym: RiSES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Principal Investigator, Maurizio Ferrarin, Dr.Eng., Ph.D., Fondazione Don Carlo Gnocchi Onlus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RISES
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-09

CONDITIONS: Stroke
Keywords: Functional Electrical Stimulation; Cerebrovascular accident; Stroke; Electromyography
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MeCFES (Experimental): 25 daily sessions (45 minutes each) of MeCFES-assisted task-oriented upper limb rehabilitation
  Interventions: Device: MeCFES-assisted task-oriented upper limb rehabilitation
- Control (Active Comparator): 25 daily sessions (45 minutes each) of usual care task-oriented upper limb rehabilitation
  Interventions: Other: Usual Care task-oriented upper limb rehabilitation

INTERVENTIONS:
Device: MeCFES-assisted task-oriented upper limb rehabilitation
  Arms: MeCFES
Other: Usual Care task-oriented upper limb rehabilitation
  Arms: Control

SUMMARY:
Goal of the present study is to evaluate the efficacy of Myoelectrically-controlled Functional Electrical Stimulation (MeCFES) for the rehabilitation of upper limb in post-stroke patients. MeCFES-assisted rehabilitation will be compared with usual care rehabilitation of upper limb. It is hypothesized that that applying MeCFES in rehabilitation to assist normal arm movements during rehabilitation of the upper limb in persons with stroke will improve the movement quality and success and thus induce recovery at the body functions level (impairment) and the activity level (disability) of the International Classification of Function (ICF) superior to that induced by usual care rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegia/hemiparesis due to a first ischemic or haemorrhagic stroke
* at least 1 month post-stroke
* willingness to participate the project
* minimum voluntary muscle activation of shoulder flexors (>1 Manual Muscle Test)
* passive Range of Motion (ROM) of the shoulder and elbow of more than 90°

Exclusion Criteria:

* epilepsy
* severe spasticity at upper limb (>= 3 Ashworth scale)
* implanted electronic device
* respiratory insufficiency
* pregnancy
* peripheral neuropathies
* cutaneous ulcers at the stimulation zone
* other use of FES on the upper limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Ferrarin, PhD, Principal Investigator — Fondazione Don Carlo Gnocchi Onlus

REFERENCES:
- [Background] van der Lee JH, Roorda LD, Beckerman H, Lankhorst GJ, Bouter LM. Improving the Action Research Arm test: a unidimensional hierarchical scale. Clin Rehabil. 2002 Sep;16(6):646-53. doi: 10.1191/0269215502cr534oa. PMID 12392340
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Wessels R, de Witte L, Andrich R, Ferrario M, Persson J, Oberg B, Oortwijn W, VanBeekum T, Lorentsen Ã. IPPA, a user-centered approach to assess effectiveness of assistive technology provision. Technol Disabil. 2000;13:105-15
- [Background] Kennedy CA, Beaton DE, Solway S, McConnell S, Bombardier C. Disabilities of the Arm, Shoulder and Hand (DASH). The DASH and QuickDASH Outcome Measure User's Manual, Third Edition. Toronto, Ontario: Institute for Work & Health, 2011.

RESULTS

PARTICIPANT FLOW:
Groups:
- MeCFES: 25 daily sessions (45 minutes each) of MeCFES-assisted task-oriented upper limb rehabilitation
  MeCFES-assisted task-oriented upper limb rehabilitation
- Control: 25 daily sessions (45 minutes each) of usual care task-oriented upper limb rehabilitation
  Usual Care task-oriented upper limb rehabilitation
Period: Overall Study
Arm/Group | MeCFES | Control
Started | 38 | 44
Completed | 32 | 36
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MeCFES | Control | Total
Number analyzed (Participants) | 38 | 44 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (12.9) | 67.1 (13.8) | 66.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 17 | 22 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change Score of ARAT Scale Between Two Time Points: Post-treatment vs Pre-treatment
Description: ARAT: Action Research Arm Test scale (15 item) (see in References section: Van der Lee JH et al 2002).
  ARAT minimum value is 0 and maximum value is 45. Higher scores mean a better outcome.
Time Frame: 5 weeks (post-treatment vs pre-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MeCFES | Control
Number analyzed (Participants) | 32 | 36
score on a scale | 6.6 (8.1) | 5.0 (7.3)

2. Primary Outcome: Change Score of FMA-UE Scale Between Two Time Points: Post-treatment vs Pre-treatment
Description: FMA-UE: Upper Extremities section of Fugl Meyer Assessment scale (see in References section: Fugl-Meyer AR et al 1975).
  FMA-UE minimum value is 0 and maximum value is 66. Higher scores mean a better outcome
Time Frame: 5 weeks (post-treatment vs pre-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MeCFES | Control
Number analyzed (Participants) | 32 | 36
score on a scale | 7.8 (9.0) | 4.5 (5.2)

3. Secondary Outcome: Change Score of IPPA Between Two Time Points: Post-treatment vs Pre-treatment
Description: IPPA: Individually Prioritized Problem Assessment (see in References section: Wessels R et al. 2000).
  IPPA minimum value is 1 and maximum value is 25. Higher scores mean worse outcome.
Time Frame: 5 weeks (post-treatment vs pre-treatment)
Population: 3 patients (1 belonging to MeCFES group and 2 to Control group) did not attend the post-treatment IPPA evaluation, thus they were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MeCFES | Control
Number analyzed (Participants) | 31 | 34
score on a scale | -2.8 (5.6) | -3.2 (3.5)

4. Secondary Outcome: Change Score of DASH Between Two Time Points: Post-treatment vs Pre-treatment
Description: DASH: Quick version of the Disability of the Arm Shoulder and Hand questionnaire (see in References section: Kennedy et al. 2011) DASH minimum value is 0 and maximum value is 100. Higher scores mean worse outcome.
Time Frame: 5 weeks (post-treatment vs pre-treatment)
Population: 2 patients (both belonging to Control group) did not attend the post-treatment DASH evaluation, thus they were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MeCFES | Control
Number analyzed (Participants) | 32 | 34
score on a scale | -4.8 (9.4) | -7.4 (11.3)

5. Secondary Outcome: Change Score of VAS for Perceived Pain Between Two Time Points: Post-treatment vs Pre-treatment
Description: VAS: Visual Analogic Scale for perceived pain on a 10-level scale. VAS minimum value is 0 and maximum value is 10. Higher scores mean worse outcome (more severe pain).
Time Frame: 5 weeks (post-treatment vs pre-treatment)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | MeCFES | Control
Number analyzed (Participants) | 32 | 36
score on a scale | 0 [-1 to 1] | 0 [-1 to 0]

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | MeCFES | Control
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/36
Other Adverse Events (participants affected / at risk) | 0/32 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes